CLINICAL TRIAL: NCT04816448
Title: Effects of Sub-Occipital Myofascial Release in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/1062
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cervicogenic Headache
Keywords: Cervicogenic headache; Pain Numerical Rating Scale; Neck disability index
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Studygroup (Experimental): cervical mobilization (Headache SNAG) with baseline treatment (Hot pack for 10 minutes, TENS 10 minutes, Neck isometrics and stretching).
  Interventions: Other: cervical mobilization (Headache SNAG)
- Control Group (Active Comparator): Sub-occipital myofascial release with baseline treatment (Hot pack for 10 minutes, TENS for 10 minutes, Neck isometrics and stretching
  Interventions: Other: Sub-occipital myofascial release

INTERVENTIONS:
Other: cervical mobilization (Headache SNAG) — For cervical mobilization the patient's position is sitting on a chair in the erect posture. The therapist handled C2 spinous process with the middle phalanx of one hand. With the other hand, he performed ventral glide asked the patient to move neck in all directions (Flexion, Extension, Side bending and rotation) one by one and then slowly move the neck back to its starting position while the therapist maintained the ventral glide.
  Arms: Studygroup
Other: Sub-occipital myofascial release — For the application of the technique , the patient position is supine lying with the head fully supported on therapist's hands and therapist places 3 middle fingers just inferior to the nuchal line, lifts the fingers tips towards the ceiling while resting the head on the table and then therapist will apply a gentle upward pull. This procedure done for 2 to 3 minutes and 5 to 7 repetitions, 3 sessions per week on alternate days were given for 6 weeks.
  Evaluation was done before treatment, during treatment at 4th week and after treatment at 6th week. Outcomes will be measured by NDI, PNRS and Universal Goniometer.
  Arms: Control Group

SUMMARY:
Cervicogenic headache is a secondary form of headache that occurs from the upper cervical spine and atlanto-occipital joint. A CGH is a frequent source of chronic headache and is frequently misdiagnosed .Cervicogenic headache is among the most common problem affecting four times more women as compared to males and is considered by some painful feeling in the head , neck ,temporal area, frontal area and around the eyes areas.

DETAILED DESCRIPTION:
There is also pain in the face and ipsilateral head that does not alternate the sides, but when cervicogenic headache becomes severe, in some patients pain may occasionally feel it on the other side of the head. Diagnosis of cervicogenic headache depends on the detailed patient's history, manual examination and the assessment of nervous system. After the diagnostic block test disappearance of headache shows that the source of this pain is cervical spine. Cervical flexion rotation test is a very useful diagnostic measure in cervical movement restriction and differential diagnosis of cervicogenic headache. Physical therapy is considered most effective treatment of cervicogenic headache in which different techniques manipulative therapy, mobilization of cervical vertebrae, stretches and sub-occipital myofascial release used.

Objective: To determine the effects of sub-occipital myofascial release in patients with cervicogenic headache.

Methods: This study was randomized control trial and on the basis of inclusion criteria, 22 patients were included and were randomized through sealed envelope in two groups A and B. Group A was given sub-occipital myofascial release along with conventional therapy while group B was given cervical mobilization and conventional therapy and both groups were assessed by using Neck Disability Index(NDI), Pain Numerical Rating Scale(PNRS) and cervical range of motion by goniometer at baseline, Week(1-4) and 8th week( last week) .The data was analyzed using SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* • Both Genders

  * Age between 20 to 75 Years
  * Neck pain referring the unilateral pain to the sub-occipital region and head.
  * Headache intensifying upon manual pressure to upper cervical joints and muscles
  * With the cranio-cervical Flexion rotation exam, neck pain and ipsilateral headache and restriction of C1 and C2 rotation.

Exclusion Criteria:

* • Tension headache (Headache on both sides)

  * If the patient not tolerate the cranio-cervical Flexion rotation test.
  * Patients presents with autonomic symptoms like visual disturbance, vertigo, dizziness.
  * If the physiotherapeutic modalities used for head pain in the last 6 months.
  * Headache other than cervical origins.
  * Clinically diagnosed as case of cervical radiculopathy or myelopathy.
  * Extreme cervical discomfort due to disk herniation, stenosis of the spinal canal and cervical arthritis.
  * Each other disorder that may be contraindicated in the upper cervical area of myofascial release.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale | 4 months
  Pain Numeric Rating Scale (PNRS) scores in subjects with moderate/severe pain at baseline. *P < 0.0001 vs. baseline. Includes only subjects with baseline PNRS score of 4 to 10. Scale ranges from 0 to 10.
NECK DISABILITY INDEX | 4 months
  the overall score range is between 0 and 50, 0 being no to little pain and discomfort while 50 being the severest degree of pain and disability with complete activity limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh LR, Chauhan V. Comparison of efficacy of myofascial release and positional release therapy in tension type headache. JMSCR. 2014;2(9):2372-9.
- [Background] Racicki S, Gerwin S, Diclaudio S, Reinmann S, Donaldson M. Conservative physical therapy management for the treatment of cervicogenic headache: a systematic review. J Man Manip Ther. 2013 May;21(2):113-24. doi: 10.1179/2042618612Y.0000000025. PMID 24421621
- [Background] Biondi DM. Cervicogenic headache: a review of diagnostic and treatment strategies. J Am Osteopath Assoc. 2005 Apr;105(4 Suppl 2):16S-22S. PMID 15928349
- [Background] Antonaci F, Sjaastad O. Cervicogenic headache: a real headache. Curr Neurol Neurosci Rep. 2011 Apr;11(2):149-55. doi: 10.1007/s11910-010-0164-9. PMID 21125430
- [Background] Fredriksen TA, Salvesen R, Stolt-Nielsen A, Sjaastad O. Cervicogenic headache: long-term postoperative follow-up. Cephalalgia. 1999 Dec;19(10):897-900. doi: 10.1046/j.1468-2982.1999.1910897.x. PMID 10668109
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743
- [Background] Bovim G, Berg R, Dale LG. Cervicogenic headache: anesthetic blockades of cervical nerves (C2-C5) and facet joint (C2/C3). Pain. 1992 Jun;49(3):315-320. doi: 10.1016/0304-3959(92)90237-6. PMID 1408296